CLINICAL TRIAL: NCT04078867
Title: Outcome of MC3 Ring Annuloplasty for Moderate and Severe Functional Tricuspid Regurgitation Associated With Rheumatic Mitral Valve Disease
Brief Title: Outcome of MC3 Ring Annuloplasty for Functional Tricuspid Regurgitation
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Yasser Ali Kamal, Principal Investigator, Minia University
Other Study IDs: 62-15
Record Dates: First submitted 2019-08-31; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Functional Tricuspid Regurgitation
Keywords: Tricuspid valve; Functional tricuspid regurgitation; Suture annuloplasty; Ring annuloplasty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- DeVega: The DeVega repair is performed when the patient had minimal annular dilation and lower severity of pulmonary hypertension
  Interventions: Procedure: tricuspid valve repair
- MC3 ring: MC3 ring annuloplasty is performed in patients with severe tricuspid annular dilation and severe pulmonary hypertension
  Interventions: Procedure: tricuspid valve repair

INTERVENTIONS:
Procedure: tricuspid valve repair — Tricuspid valve repair during mitral valve replacement for rheumatic heart disease using suture (DeVega) repair or ring annuloplasty

SUMMARY:
This study includes 105 patients who underwent repair for ≥ moderate tricuspid regurgitation (TR) during mitral valve replacement for rheumatic valve disease. Between January 2016 and December 2018, a group of 23 patients underwent ring annuloplasty with Edward MC3 rings were compared to another group of 82 patients underwent standard suture (DeVega) repair. The primary outcome was residual TR (≥ moderate TR).

DETAILED DESCRIPTION:
This study evaluated early and midterm outcomes after operations for TV repair which were performed at our institution, between January 2016 and December 2018. The mean follow-up duration was 18.84±9.90 months (range: 3-33 months). The study included 105 patients who underwent repair for FTR during mitral valve replacement for rheumatic valve disease. There were 82 patients underwent suture (DeVega) repair and 23 patients underwent ring annuloplasty using Edward MC3 incomplete 3D ring. The indications of surgery for FTR were: (1) severe TR; or (2) moderate TR with annular dilatation greater than 40 mm and/or preoperative systolic pulmonary artery pressure (SPAP) >50 mmHg. We excluded patients with non-rheumatic mitral disease, combined mitral and aortic valve replacement, mitral valve repair, concomitant coronary artery or aortic surgery, mild or organic tricuspid regurgitation, emergency surgery, reoperations or missed data. Based on echocardiographic data, the severity of TR was graded as: 0 (no TR), 1+ (mild TR), 2+ (mild to moderate TR), 3+ (moderately severe TR), or 4+ (severe).

The type of tricuspid valve repair was chosen in according to surgeon's preference and echocardiographic criteria of TV. The DeVega repair was performed when the patient had minimal annular dilation and lower severity of pulmonary hypertension, while ring annuloplasty was performed in patients with severe tricuspid annular dilation and severe pulmonary hypertension. The DeVega repair was performed on a beating heart using pledget-supported two 4-0 polypropylene running parallel sutures. The MC3 ring annuloplasty was performed through right atriotomy using cardiopulmonary bypass and cardioplegic arrest. The ring size was determined after measurement of the length of the attachments of the tricuspid septal leaflet (the distance between the anteroseptal and septoposterior commissures) or the surface area of the anterior leaflet. The chosen ring was undersized by at least one size. The ring was implanted from the anteroseptal commissure to the middle of the septal leaflet. A series of 8 to10 mattress sutures with a 2-0 Ethibond multifilament suture were made on the tricuspid annulus starting from the center of the septal annulus to the anteroseptal commissure in the counter-clockwise direction, to avoid the atrioventricular conduction tissue. Thereafter, the sutures were placed through the sewing ring of the prosthesis , followed by lowering and securing of the ring to the annulus The collected pre-operative data included age, sex, New York Heart Association (NYHA) functional class, , and the type of preoperative mitral valve disease. The primarily assessed post-operative outcome was residual TR (≥ moderate TR; ≥ grade +2). Other assessed pre- and post-operative parameters included NYHA functional class, and echocardiographic data regarding grade of TR, SPAP, tricuspid annulus (TA) diameter, tricuspid annular plane systolic excursion (TAPSE), left atrial diameter (LAD), left ventricular end-diastolic dimension (LVEDD), left ventricular end-systolic dimension (LVESD), and left ventricular ejection fraction (LVEF).

ELIGIBILITY:
Inclusion Criteria:

* Rheumatic mitral valve disease
* Surgery for mitral valve replacement
* Severe functional tricuspid regurgitation
* Moderate functional tricuspid regurgitation with annular dilatation > 40 mm
* Moderate functional tricuspid regurgitation with preoperative systolic pulmonary artery pressure (SPAP) >50 mmHg

Exclusion Criteria:

* Patients with non-rheumatic mitral disease
* Combined mitral and aortic valve replacement
* Mitral valve repair
* Concomitant coronary artery or aortic surgery
* Mild or organic tricuspid regurgitation
* Emergency surgery
* Reoperations
* Invalid or missed data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent repair for functional tricuspid regurgitation during mitral valve replacement for rheumatic valve disease
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Residual tricuspid regirgitation (TR) | 3-33 months
  residual TR is defined when there is moderate or above degree of TR at the last follow-up echocardiography of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Yasser A Kamal, MD, Principal Investigator — Minia University

IPD SHARING:
Plan to Share IPD: Undecided